CLINICAL TRIAL: NCT02805777
Title: Long Term Vent Flow Study of Prototype Nasal CPAP Mask System
Brief Title: Vent Flow Study of Prototype Nasal CPAP Mask
Acronym: GVFECT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study not required due to change in device
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA300516
Record Dates: First submitted 2016-06-01; First posted 2016-06-20 (Estimated); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Obstructive Sleep Apnea (OSA)
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Washing procedure 1 (Experimental): this group will apply washing technique 1
  Interventions: Device: CPAP mask
- Washing procedure 2 (Experimental): this group will apply washing technique 2
  Interventions: Device: CPAP mask

INTERVENTIONS:
Device: CPAP mask — A new vent CPAP mask system will be used in this trial

SUMMARY:
As continuous positive airway pressure is the treatment choice for OSA, a mask is vital in ensuring the effectiveness of therapy delivery. The study will evaluate the performance of a new mask system with diffuse vent technology. This is done by characterizing the mask flow over time and compare the performance between patients who apply 2 different washing procedures to the mask. The study will also subjectively assess breathing comfort and performance of the mask system.

ELIGIBILITY:
Inclusion Criteria:

* Participants willing to give written informed consent
* Participants who can read and comprehend English
* Participants using APAP for >6 months
* Participants who are willing to use the mask system for the 3 month duration of the trial.
* Participants who are over 18 years of age
* Participants who currently use a nasal mask system

Exclusion Criteria:

* Participants not willing to give written informed consent
* Participants who cannot read and comprehend English
* Participants using an inappropriate mask system
* Participants on a Bilevel or ASV therapy
* Participants who are pregnant
* Participants with a pre-existing lung disease/ condition that would predispose them to pneumothorax (for example: COPD, lung cancer lung injury; fibrosis of the lungs; recent (< 2years) case of pneumonia or lung infection
* Participants or whose bed partner with implantable metallic implants in the head, neck and chest region affected by magmetic fields (Non-ferrous implants may be acceptable)
* Participants that weight <30 kg
* Participants who are unsuitable to participate in the study in the opinion of the researcher

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05-01 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Changes in vent flow of the mask system, which will be recorded on a flow testing rig (units= LPM). Baseline flow in LPM will be compared to that at the conclusion of the trial. | 12 weeks
  The mask system will be flow tested after use when returned by the participant at each scheduled visit. The flow of the mask system will be recorded as per the mask to flow procedure of ISO17510 Sleep apnoea breathing therapy - Part 2: Annex B Exhaust flow test procedure.
  The results will be reported as an average flow in LPM. Results will be presented graphically with average flow on the vertical axis and use time (weeks) on the horizontal axis. This will allow us to assess any changes in vent flow over time.

SECONDARY OUTCOMES:
Parameters such as the apnoea/hypopnoea index (AHI) will be recorded and analysed | 12 weeks
Questionnaire to assess the perceived overall performance of the mask by the participant. Questions around comfort will be asked. | 12 weeks
  This data will be collected from questionnaires completed in the home environment during use of the mask. The outcome will be descriptive in nature. When there is a single rating which expresses how good the product is, we will set a criterion value C which will be regarded as acceptable. The statistical test used will be the Wilcoxon signed ranks method.
Bioburden quantification by laboratory testing of venting components at end of trial | 12 weeks
  The viable microorganisms present on the mask system upon completion of the trial will be counted using ISO 11737 Sterilisation of medical devices - Microbiological methods - Part 1: Determination of a population of microorganisms on products.
  Results will be presented as total quantity of Microorganism (log10 CFU) per diffuser.

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Schindhelm, PhD, Principal Investigator — ResMed/The University of New South Wales

IPD SHARING:
Plan to Share IPD: No
There is no sharing plan.